CLINICAL TRIAL: NCT07356830
Title: Effect of Music Therapy on Psychological State and Pregnancy Outcome of Patients With Artificial Insemination
Brief Title: Nurse-Led Staged Art Therapy Effects on Psychological Distress and Pregnancy Outcomes in AIH: RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KY-2025-193
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Music Therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group : on the basis of the control group with music therapy. (Experimental): on the basis of the control group with music therapy.
  Interventions: Other: music therapy

INTERVENTIONS:
Other: music therapy — Experimental group : on the basis of the control group with music therapy.

SUMMARY:
Music therapy is a comprehensive therapy that integrates musicology, psychology and medicine. It is an application and development outside the field of traditional art appreciation and aesthetics . Clinical studies have shown that music therapy can improve the patient 's sense of tension, relieve anxiety, and has a certain effect of auxiliary analgesia. At the same time, music therapy is easy to operate, economical and feasible, non-invasive and safe , and improves physical and mental health. Music therapy can work through the hypothalamus-pituitary and other multi-system cross-activity, arouse the patient 's pleasant thoughts and emotional experience, and has the function of regulating psychology and physiology . Many studies at home and abroad have shown that most infertility patients have negative emotions, such as anxiety and depression For Chinese women, affected by the traditional culture of " no filial piety, no filial piety, no filial piety, " patients are under greater reproductive pressure. Many studies have confirmed that psychological stress can affect the function of the hypothalamus-pituitary-ovarian axis, inhibit the secretion of gonadotropins by the pituitary gland, interfere with follicular growth, affect the developmental potential of oocytes and embryos, and thus affect reproductive function . Psychological stress can also interfere with embryo implantation by inhibiting endometrial receptivity . Anxiety can promote sympathetic nerve excitation, release more catecholamines, hinder the growth of follicles in the ovary and the secretion of luteinizing hormone, and affect the clinical effect of superovulation. The decrease of estrogen and progesterone secretion affects the number and quality of follicles and the development of endometrium, thus reducing the pregnancy rate Long-term depression can also endanger physical health, destroy pregnancy outcomes, and lead to abortion. With the development of medicine, the ' biological-psychological-social ' medical model has been paid more and more attention, and the psychological factors in the treatment of infertility have also attracted more and more attention. Although the mechanism of music therapy is not yet clear, studies have shown that it can inhibit the secretion of endogenous hormones such as adrenaline.

ELIGIBILITY:
Inclusion Criteria:①aged 20-40 years old, conscious, with normal language expression ability and understanding ability ;②Exclusion of mental illness and serious diseases of vital organs, voluntary participation in the survey. ③ Patients who met the WHO diagnostic criteria for infertility : those who had normal sexual life after marriage without contraception for 1 year or more.

Exclusion Criteria:①Those who could not cooperate with the scale due to deafness, dumbness, aphasia and disturbance of consciousness ; ② patients with mental disorders and severe important organ diseases.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 254 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | Pregnant was checked 14 days after the end of artificial insemination.
  Pregnant was checked 14 days after the end of artificial insemination.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fouth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes